CLINICAL TRIAL: NCT03140397
Title: Examination of the Bioavailability and Bioactivity of the Two Natural Food Ingredients 6-Prenylnaringenin and 8-Prenylnaringenin.
Brief Title: Oral Bioavailability and Bioactivity of Prenylflavonoids From Hops
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Hohenheim (Other)
Collaborators: Universität Tübingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HS-PF1-2016
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Safety After Oral Intake; Pharmacokinetics After Oral Intake; Immune Cells Activity
Keywords: Bioavailability; Pharmacokinetics; 8-prenylnaringenin; 6-prenylnaringenin; Prenylflavonoids; PBMC
MeSH Terms: interventions — 6-prenylnaringenin; 8-prenylnaringenin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Capsules filled with mannitol and silicon dioxide
  Interventions: Dietary Supplement: Placebo
- 6-prenylnaringenin (Experimental): 500 mg 6-PN plus mannitol and silicon dioxide
  Interventions: Dietary Supplement: 6-prenylnaringenin
- 8-prenylnaringenin (Experimental): 500 mg 8-PN plus mannitol and silicon dioxide
  Interventions: Dietary Supplement: 8-prenylnaringenin

INTERVENTIONS:
Dietary Supplement: Placebo
  Arms: Placebo
Dietary Supplement: 6-prenylnaringenin
  Other Names: 6-PN
  Arms: 6-prenylnaringenin
Dietary Supplement: 8-prenylnaringenin
  Other Names: 8-PN
  Arms: 8-prenylnaringenin

SUMMARY:
The prenylflavonoids 6-prenylnaringenin (6-PN) and 8-prenylnaringenin (8-PN) are secondary plant substances, almost exclusively found in hops (Humulus lupulus). Both compounds have known potential biological properties, but poor bioavailability due to their low oral absorption and retention. Our study followed a single dose (500 mg 6- or 8-PN), placebo controlled, randomized, double-blind, three armed crossover study design with ≥2-week washout periods. Plasma, PBMC and urine samples were collected at intervals up to 24 h after intake. Investigators investigated the safety, pharmacokinetics and impact of oral prenylflavonoids on the function of cells of the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers with blood chemistry values within normal ranges
* Age: 18-45 years
* BMI: 19-25 kg/m2

Exclusion Criteria:

* Pregnancy or lactation
* Alcohol and/or drug abuse
* Use of dietary supplements or any medications, except contraceptives
* Any known malignant, metabolic and endocrine diseases
* Previous cardiac infarction
* Dementia
* Participation in a clinical trial within the past 6 weeks prior to recruitment
* Physical activity of more than 5 h/wk

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-01; Primary Completion 2017-04 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Mean area under the curve (AUC) of plasma concentration vs. time of total 6-prenylnaringenin [nmol/L*h] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
  Total 6-PN after deconjugation with beta-glucuronidase/sulphatase
Mean area under the curve (AUC) of plasma concentration vs. time of total 8-prenylnaringenin [nmol/L*h] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
  Total trans-epsilon-viniferin after deconjugation with beta-glucuronidase/sulphatase
Mean maximum plasma concentration (Cmax) of total 6-prenylnaringenin [nmol/L] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
  Total trans-resveratrol after deconjugation with beta-glucuronidase/sulphatase
Mean maximum plasma concentration (Cmax) of total 8-prenylnaringenin [nmol/L] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
  Total trans-epsilon-viniferin after deconjugation with beta-glucuronidase/sulphatase
Time to reach maximum plasma concentration (Tmax) of total 6-prenylnaringenin [h] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
  Total trans-resveratrol after deconjugation with beta-glucuronidase/sulphatase
Time to reach maximum plasma concentration (Tmax) of total 8-prenylnaringenin [h] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
  Total trans-epsilon-viniferin after deconjugation with beta-glucuronidase/sulphatase
Cumulative urinary excretion of total 6-prenylnaringenin [nmol/g creatinine] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
  Total trans-resveratrol after deconjugation with beta-glucuronidase/sulphatase
Cumulative urinary excretion of total 8-prenylnaringenin [nmol/g creatinine] | 0, 0.5, 1, 2, 4, 6, 8 and 24 h post dose
  Total trans-epsilon-viniferin after deconjugation with beta-glucuronidase/sulphatase
Cell count (dead cells/ml and living cells/ml) of PBMCs after 6-PN administration | 0, 6, and 24 h post dose
Cell count (dead cells/ml and living cells/ml) of PBMCs after 8-PN administration | 0, 6, and 24 h post dose
Cell viability of PBMCs after 6-PN administration | 0, 6, and 24 h post dose
Cell viability of PBMCs after 8-PN administration | 0, 6, and 24 h post dose

SECONDARY OUTCOMES:
Serum aspartate transaminase activity [U/L] | 0, 4, 24h post-dose
Serum alanine transaminase activity [U/L] | 0, 4, 24h post-dose
Serum gamma-glutamyl transferase activity [U/L] | 0, 4, 24h post-dose
Serum alkaline phosphatase activity [U/L] | 0, 4, 24h post-dose
Serum bilirubin | 0, 4, 24h post-dose
Serum uric acid [mg/dL] | 0, 4, 24h post-dose
Serum creatinine [mg/dL] | 0, 4, 24h post-dose
Serum total cholesterol [mg/dL] | 0, 4, 24h post-dose
Serum HDL cholesterol [mg/dL] | 0, 4, 24h post-dose
Serum LDL cholesterol [mg/dL] | 0, 4, 24h post-dose
Serum triacylglycerols [mg/dL] | 0, 4, 24h post-dose
LDL/HDL cholesterol ratio | 0, 4, 24h post-dose
Serum cystatin C [mg/mL] | 0, 4, 24h post-dose
Glomerular filtration rate [mL/min] | 0, 4, 24h post-dose
Serum glucose [mg/dL] | 0, 24h post-dose
Hemoglobin [g/dL] | 0, 24h post-dose
Mean corpuscular hemoglobin concentration [g/dL] | 0, 24h post-dose
Mean corpuscular hemoglobin [pg] | 0, 24h post-dose
Mean corpuscular volume [fL] | 0, 24h post-dose
Hematocrit [%] | 0, 24h post-dose
Erythrocytes [/pL] | 0, 24h post-dose
Thrombocytes [/nL] | 0, 24h post-dose
Leucocytes [/nL] | 0, 24h post-dose
Segmented granulocytes [%] | 0, 24h post-dose
Lymphocytes [%] | 0, 24h post-dose
Monocytes [%] | 0, 24h post-dose
Basophil granulocytes [%] | 0, 24h post-dose
Eosinophil granulocytes [%] | 0, 24h post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Jan Frank, Prof. Dr., Principal Investigator — University of Hohenheim; Sascha Venturelli, Dr. med. Dr. rer. nat., Principal Investigator — Eberhard Karls University Tuebingen; Christian Busch, Dr. med., Principal Investigator — Eberhard Karls University Tuebingen
Locations (2):
- Germany (2):
  - University of Hohenheim, Stuttgart, Baden-Wurttemberg
  - Eberhard Karls University Tuebingen, Tübingen, Baden-Wurttemberg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Calvo-Castro LA, Burkard M, Sus N, Scheubeck G, Leischner C, Lauer UM, Bosy-Westphal A, Hund V, Busch C, Venturelli S, Frank J. The Oral Bioavailability of 8-Prenylnaringenin from Hops (Humulus Lupulus L.) in Healthy Women and Men is Significantly Higher than that of its Positional Isomer 6-Prenylnaringenin in a Randomized Crossover Trial. Mol Nutr Food Res. 2018 Apr;62(7):e1700838. doi: 10.1002/mnfr.201700838. Epub 2018 Mar 1. PMID 29363261
- See also: Website of the research group — http://www.nutrition-research.de/